CLINICAL TRIAL: NCT05464576
Title: Tumor Staging T of Bladder Tumours: Correlation of MRI and Anatomopathologic Analysis.
Acronym: IRMAA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AOI 2021 GUY; 2022-A00400-43 (Other: CHU Gabriel MONTPIED - CLERMONT FERRAND)
Record Dates: First submitted 2022-07-12; First posted 2022-07-19 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-07

CONDITIONS: Urinary Bladder Tumour; MRI; Invasion; Diagnosis
Keywords: Magnetic resonance imaging; MRI versus anatomopathology; Urinary bladder tumor; MRI diagnosis before TURB (Trans Urethral Resection of the Bladder); NIMBC (Non Invasive Muscle Bladder Cancer)
MeSH Terms: conditions — Disease; Urinary Bladder Neoplasms; Non-Muscle Invasive Bladder Neoplasms

STUDY DESIGN:
Intervention Model Description: All participants receive the same intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Comparison between MRI versus anatomopathology report in bladder cancer (Other): Comparison of MRI and anatomopathology on urinary bladder tumour after transurethral resection of the bladder or cystectomy (for patients with an invasive bladder cancer.
  Interventions: Diagnostic Test: MRI

INTERVENTIONS:
Diagnostic Test: MRI — Using the MRI in the diagnosis of the bladder cancer (invasive or not)

SUMMARY:
Urinary bladder tumors with a frequency of 13000 new cases a year, have a heterogeneity in terms of survival according to the stage of local flooding.

This is an aggressive tumor because of the potential muscular infiltration. It seems important in this case (muscular invasion), to increase the global survival.

The anatomopathological analysis of the TURB (biopsy byTrans-Urethral Resection of the Bladder) is actually the gold standard for the pathology of bladder tumor.

No need an imaging to discuss about the small and non muscular invasive tumor. But in most cases, the use is to perform at last an ultrasound or a CT-Scan, specially for the invasive tumor.

A lot of studies show that CT SCAN. is not the best way of investigation for the bladder muscle invasion. However, as in the prostate cancer with the PIRADS Score, the MRI can be useful for the bladder, thanks to the sequence improvement to the machine.

The study from Panebianco 2018, starts to talk about the MRI in the urinary bladder cancer with new radiological terms. It creates a new score called VIRADS score (as the PIRADS score already used for the prostate cancer). But it is never compared with the results of the TURB.

Our study compares the results of the MRI pre operative versus the pathology results on prospective analysis.

Main objective : T tumoral score in urinary bladder tumor : MRI versus pathology results.

Secondary objectives : the contribution of diffusion weighted MRI in the bladder neoplasm.

Type of study : interventional study, prospective, mono centric, single arm, intent-to-treat

DETAILED DESCRIPTION:
This is a single center study comparing MRI report to anatomopathological report in participants who were diagnosed with an urinary bladder tumour, histologically confirmed in routine care.

Bladder tumours are frequent pathologies with 13,000 new cases per year in France. They can present various types of damage, from the most benign to the most serious stages, depending on the number, the extent of the lesions and their degree of infiltration (superficial or deeper). We also know that the shorter the treatment time, the better the final prognosis. An infiltrating lesion taken as soon as it is discovered considerably reduces the likelihood of progression. It is therefore necessary to improve patient care.

Currently, when a bladder lesion is visualized by the urologist during the cystoscopy (examination during which the urologist notes the presence or absence of bladder lesion(s)), the only way to know its stage (and its degree of infiltration if applicable) which will determine the follow-up care, consists in carrying out an intervention called Trans Urethral Resection of the Bladder (TURB), in order to remove the lesions which will be analyzed in the anatomopathological laboratory. This analysis is the best interpretation of the tumour stage, carried out in accordance with the international standards, and the only way to have a diagnosis of tumour lesions. Indeed, to date, no imaging technique (ultrasound, scanner, etc.) makes it possible to obtain it.

The CT scan of the urinary tract is currently only used to identify lesions of the upper urinary tract or lymph nodes.

However, in recent years, these techniques have evolved considerably, and studies have shown that MRI seems to have the ability to determine the tumour stage of bladder lesions.

Investigators propose to demonstrate the value of MRI in determining tumour infiltration compared to the anatomopathological analysis of samples taken during TURB. This would provide better patient care in human, pathological, economic and technical terms, by developing a more precise mapping of lesions in the bladder, reducing waiting times for results and therefore obtaining earlier diagnosis, a reduction in the number of consultations, hospitalizations, surgeries more or less morbid, examinations...

Finally, this would potentially :

* Reduce the number of cystoscopies (examination normally painless, but unpleasant and frequent) carried out before TURB but also throughout the monitoring following the TURB,
* Detect very early infiltrating lesions in order to limit their potential extension before the cystectomy.

ELIGIBILITY:
Inclusion Criteria:

* Patient, male or female, aged >18ans
* Benefiting from Social Security
* Urinary bladder tumour confirmed on cystoscopy and requiring a TURB
* Understanding and reading French well
* Ability to give informed consent

Exclusion Criteria:

* Participation refusal
* MRI contraindication : pacemaker, heart valve, clips, stents, coils, non-MRI compatible defibrillators, neural or peripheral stimulator, cochlear implant, intraocular foreign body, claustrophobia
* Patient under guardianship, deprived of liberty, impaired understanding
* Pregnant/breastfeeding woman
* Allergy to gadolinium (contrast product necessary for carrying out the MRI), hypersensitivity to gadoteric acid or gadolinated contrast products, to meglumine
* Suspicion of an infectious disease such as schistosomiasis (differential diagnosis)
* Patient presenting with macroscopic clotting hematuria on the day of the MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Non inferiority of the MRI compared to TURB in determining the degree of tumour infiltration | through study completion, up to 6 month
  Compare the concordance between MRI and pathological analysis of the samples of the TURB in determining the degree of bladder tumour infiltration.
  The dependent variable of interest is the determination of the infiltrating character (or not) of the tumour on the anatomopathological examination of the RTUV. It will be confronted with the main explanatory variable, which is the determination of the invasive character (or not) of the tumour on the preoperative MRI.

SECONDARY OUTCOMES:
Non inferiority of MRI versus anatomopathological report of the cystectomy | through study completion, an average of 6 month
  Compare the concordance between MRI and pathological analysis of the cystectomy on the presence or absence of tumour residue after neoadjuvant chemotherapy.
  The dependent variable of interest is the determination of the presence (or not) of a tumour on the anatomopathological examination of the cystectomy. It will be confronted with the main explanatory variable, which is the determination of the presence (or not) of tumour on the post neoadjuvant chemotherapy MRI.
Efficacy of neoadjuvant chemotherapy on muscle invasive bladder tumour | through study completion, an average of 6 month
  Determine the number of cystectomy parts without tumour residue after neoadjuvant chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Laurent GUY, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU clermont-ferrand, Clermont-Ferrand, France